CLINICAL TRIAL: NCT00295750
Title: An Open-label, Multi-Centre, Randomized, Parallel-group Study, Investigating the Efficacy and Safety of Degarelix One Month Dosing Regimens; 160 mg (40 mg/ml) and 80 mg (20mg/ml), in Comparison to LUPRON DEPOT® 7.5 mg in Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: The Efficacy and Safety of Degarelix One Month Dosing Regimens in Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS21
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Results first posted 2009-04-16 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- degarelix 240/160 mg (Experimental): Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 160 mg SC (by injection under the skin) given every 28 days.
  Interventions: Drug: Degarelix
- degarelix 240/80 mg (Experimental): Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 80 mg SC (by injection under the skin) given every 28 days.
  Interventions: Drug: Degarelix
- Leuprolide 7.5 mg (Active Comparator): Leuprolide (Lupron Depot) 7.5 mg IM (in the muscle) every 28 days starting at day 0.
  Interventions: Drug: Leuprolide 7.5 mg

INTERVENTIONS:
Drug: Degarelix — Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 160 mg SC (by injection under the skin) given every 28 days for 364 days.
  Other Names: FE200486
  Arms: degarelix 240/160 mg
Drug: Degarelix — Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 80 mg SC (by injection under the skin) given every 28 days for 364 days.
  Other Names: FE 200486
  Arms: degarelix 240/80 mg
Drug: Leuprolide 7.5 mg — Leuprolide (Lupron Depot) 7.5mg IM (in the muscle every 28 days starting at day 0.
  Other Names: Lupron
  Arms: Leuprolide 7.5 mg

SUMMARY:
The study was a three-arm, active-control, multi-centre, parallel group study.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients, aged 18 years or over, with histologically proven prostate cancer of all stages in whom endocrine treatment is indicated.
* Baseline testosterone >1.5 ng/mL.
* Life expectancy of at least 12 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (35):
- United States (23):
  - Urology Centers of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Advanced Urology Medical Center, Anaheim, California
  - Pacific Clinical Center, Beverly Hills, California
  - Simi-San Faernando Valley Urology Associates, Granada Hills, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - Western Clinical Research, Torrance, California
  - Urology Associate PC, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Regional Urology, Shreveport, Louisiana
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Jay A. Motola, MD, FACS, Carmel, New York
  - Northeast Urology Research, Concord, North Carolina
  - The Urology Center, Greensboro, North Carolina
  - State College Urologic Association, State College, Pennsylvania
  - Univeristy Urological Research Institute, Providence, Rhode Island
  - University Urological Research Institute, Providence, Rhode Island
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology San Antonio Research, San Antonio, Texas
  - Urology of Virginia Research, Norfolk, Virginia
  - Office of Jeffrey Frankel, Seattle, Washington
- Bruce W. Palmer Urology Inc, 125-70 Exhibition Street, Kentville, Nova Scotia, Canada
- Nemocnice Jindrichuv Hradec a.s., U Nemocnice 380/III, Jindřichův Hradec, Czechia
- Urologische Klinik, Universitatsklinikum Mannheim, Theodor-Kutzer-Ufer 1-3, Mannheim, Germany
- Szeged M.J.V.O. Korhaza, Urologiai Osztaly, Kalvaria sugarut 57, Szeged, Hungary
- Hospital General "Dr Santiago Ramon y Cajal", ISSSTE, Predio Canoas S/N, Durango, DGO, Mexico
- Atrium MC, Henri Dunantstraat 5, Heerlen, Netherlands
- Puerto Rico (2):
  - Cristo Redentor Hospital, La Hacienda
  - San Juan VA Medical Center, San Juan
- Provita Center, 2 Primaverii Street, Constanța, Romania
- Andros Urology Clinic, Ulitsa Lenina 36A, Saint Petersburg, Russia
- Kiev City Clinical Hospital #3, Petr Ivaschenko 26, Petra Zaporogtsa str., Kiev, Ukraine
- Derriford Hospital, Derriford Road, Plymouth, United Kingdom

REFERENCES:
- [Result] Klotz L, Boccon-Gibod L, Shore ND, Andreou C, Persson BE, Cantor P, Jensen JK, Olesen TK, Schroder FH. The efficacy and safety of degarelix: a 12-month, comparative, randomized, open-label, parallel-group phase III study in patients with prostate cancer. BJU Int. 2008 Dec;102(11):1531-8. doi: 10.1111/j.1464-410X.2008.08183.x. PMID 19035858
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Groups:
- Leuprolide 7.5 mg: Lupron Depot 7.5 mg IM (in the muscle) every 28 days starting at day 0.
Period: Overall Study
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Started | 206 (randomized) | 210 (randomized) | 204 (randomized)
Intent-to-treat (ITT) Population | 202 (randomized and exposed patients) | 207 (randomized and exposed patients) | 201 (randomized and exposed patients)
Completed | 163 | 169 | 172
Not Completed | 43 | 41 | 32
Not completed — Adverse Event | 19 | 15 | 12
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Taking prohibited therapy | 2 | 3 | 2
Not completed — Administrative errors | 2 | 4 | 5
Not completed — Trial drug errors | 1 | 1 | 0
Not completed — Disease progression | 2 | 1 | 0
Not completed — Personal reasons | 0 | 1 | 0
Not completed — Randomized but never received trial drug | 4 | 3 | 3
Not completed — Withdrawal by Subject | 9 | 4 | 7
Not completed — Protocol Violation | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg | Total
Number analyzed (Participants) | 202 | 207 | 201 | 610
Age, Categorical [Count of Participants; unit: Participants] — Intent-to-treat (ITT) population.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 37 | 43 | 38 | 118
    >=65 years | 165 | 164 | 163 | 492
Age Continuous [Median (Full Range); unit: years] — ITT population.
  years | 72 (8.47) [50 to 88] | 72 (8.12) [51 to 89] | 74 (8.77) [52 to 98] | 73 (8.45) [50 to 98]
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population.
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 202 | 207 | 201 | 610
Race (NIH/OMB) [Count of Participants; unit: Participants] — ITT population
  Participants
    American Indian or Alaska Native | 22 | 18 | 19 | 59
    Asian | 1 | 1 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 11 | 17 | 10 | 38
    White | 168 | 171 | 172 | 511
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — ITT population
  participants
    North America | 84 | 87 | 86 | 257
    Europe | 118 | 120 | 115 | 353
Curative Intent [Number; unit: participants] — ITT population. Curative intent refers to radical prostatectomy or radiotherapy.
  participants
    Yes | 24 | 30 | 24 | 78
    No | 178 | 177 | 177 | 532
Gleason Score [Number; unit: participants] — ITT population. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive. Gleason scores were unavailable for 3 patients.
  participants
    2-4 | 21 | 20 | 24 | 65
    5-6 | 67 | 68 | 63 | 198
    7 | 56 | 63 | 62 | 181
    8-10 | 56 | 56 | 51 | 163
Stage of Prostate Cancer [Number; unit: participants] — ITT population. Stage of prostate cancer was classified according to the Tumour, Nodule and Metastatic classification that is a cancer staging system that describes the extent of cancer. T describes the size of the tumor and whether it has invaded nearby tissue, N describes regional lymph nodes that are involved, and M describes distant metastasis
  participants
    Localized | 59 | 69 | 63 | 191
    Locally advanced | 62 | 64 | 52 | 178
    Metastatic | 41 | 37 | 47 | 125
    Not classifiable | 40 | 37 | 39 | 116
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — ITT population
  kilogram per square meter | 26.6 (3.70) | 26.7 (4.21) | 26.9 (3.86) | 26.8 (3.93)
Serum Prostate-specific Antigen Levels [Median (Inter-Quartile Range); unit: nanogram per milliliter] | 19.9 [8.2 to 68] | 19.8 [9.4 to 46] | 19.0 [8.7 to 57] | 19.0 [8.7 to 57]
Serum Testosterone Levels [Median (Inter-Quartile Range); unit: nanogram per milliliter] | 3.78 [2.86 to 5.05] | 4.11 [3.05 to 5.32] | 3.84 [2.91 to 5.01] | 3.93 [2.89 to 5.10]
Time Since Prostate Cancer Diagnosis [Mean (Standard Deviation); unit: days] — ITT population.
  days | 485 (1109) | 491 (994) | 497 (1088) | 491 (1063)
Weight [Mean (Standard Deviation); unit: kilogram] — ITT population
  kilogram | 78.7 (13.0) | 79.8 (14.9) | 79.4 (12.2) | 79.3 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Testosterone <=0.5ng/mL From Day 28 Through Day 364
Description: Kaplan-Maier estimates of the cumulative probabilities of testosterone <=0.5 ng/mL from Day 28 to Day 364. The degarelix response rate estimation determined whether the lower bound of the 95% confidence interval for the cumulative probability of testosterone <=0.5 ng/mL from Day 28 to Day 364 was no lower than 90%.
Time Frame: 12 months
Population: Intent-to-treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
percentage of patients | 98.3 [94.8 to 99.4] | 97.2 [93.5 to 98.8] | 96.4 [92.5 to 98.2]
Statistical Analysis 1: Comparison: Degarelix 240/160 mg vs Leuprolide 7.5 mg; A non-inferiority assessment determined whether degarelix was non-inferior to leuprolide with respect to the cumulative probability of testosterone <=0.5 ng/mL from Day 28 to Day 364; Test type: Non-Inferiority or Equivalence — The non-inferiority limit was -10 percentage points; Difference in cumulative probability = 1.9, 97.5% CI [-1.8 to 5.7]
Statistical Analysis 2: Comparison: Degarelix 240/80 mg vs Leuprolide 7.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority limit was -10 percentage points; Difference in cumulative probability = 0.9, 97.5% CI [-3.2 to 5.0]

2. Secondary Outcome: Percentage of Patients With Testosterone Surge During the First Two Weeks of Treatment
Description: A patient was defined as having a testosterone surge if the testosterone level exceeded baseline by >=15% on any two days during the first two weeks of treatment (i.e. two of Study Days 1, 3, 7 and 14).
Time Frame: 2 weeks
Population: ITT population. If one or more of the testosterone values on Days 1, 3, 7 or 14 was missing, the last observation was carried forward.
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
percentage of patients | 0.5 [0.0 to 2.7] | 0.0 [0.0 to 1.8] | 80.1 [73.9 to 85.4]
Statistical Analysis 1: Comparison: Degarelix 240/160 mg vs Leuprolide 7.5 mg; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Degarelix 240/80 mg vs Leuprolide 7.5 mg; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Percentage of Patients With Testosterone Level <=0.5 ng/mL at Day 3
Description: This outcome measure presents the testosterone levels 3 days after the initial dose of trial medication.
Time Frame: 3 days
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
percentage of patients | 95.5 [91.7 to 97.9] | 96.1 [92.5 to 98.3] | 0 [0 to 1.8]
Statistical Analysis 1: Comparison: Degarelix 240/160 mg vs Leuprolide 7.5 mg; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Degarelix 240/80 mg vs Leuprolide 7.5 mg; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Frequency and Size of Testosterone Changes at Day 255 and/or Day 259 Compared to the Testosterone Level at Day 252
Description: Testosterone increases on Day 255 and/or on Day 259 (highest value of Day 255 and Day 259 was used) were compared with Day 252 values. Patients were categorised with shifts of <=-0.25, >-0.25-0, >0-0.25, >0.25-0.5 and >0.5 ng/mL from mean testosterone levels on Day 252.
Time Frame: Day 252, Day 255, and Day 259
Population: ITT population who had blood samples drawn on Day 252, Day 255, and Day 259.
Measure: Number; unit: participants
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 176 | 178 | 179
participants
  <=-0.25 ng/mL | 1 | 3 | 0
  >-0.25-0 ng/mL | 84 | 85 | 49
  >0-0.25 ng/mL | 91 | 90 | 122
  >0.25-0.5 ng/mL | 0 | 0 | 5
  >0.5 ng/mL | 0 | 0 | 3

5. Secondary Outcome: Percentage Change in Prostate-specific Antigen From Baseline to Day 14 and Day 28
Description: Percentage change from Baseline to Day 14 and Day 28 in prostate-specific antigen, which is a clinically important biological marker for treatment effect and prostate cancer progression.
Time Frame: Days 14 and 28
Population: ITT population.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
percent change
  Day 14 | -64.6 [-77.8 to -40.8] | -63.4 [-77.1 to -48.4] | -17.9 [-35.5 to -5.2]
  Day 28 | -82.3 [-91.4 to -68.3] | -84.9 [-91.6 to -73.2] | -66.7 [-81.3 to -47.7]
Statistical Analysis 1: Comparison: Degarelix 240/160 mg vs Leuprolide 7.5 mg; Percentage change from baseline to Day 14; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Degarelix 240/80 mg vs Leuprolide 7.5 mg; Percentage change from baseline to Day 14; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Degarelix 240/160 mg vs Leuprolide 7.5 mg; Percentage change from baseline to Day 28; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Degarelix 240/80 mg vs Leuprolide 7.5 mg; Percentage change from baseline to Day 28; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Participants Grouped by Time to Prostate-specific Antigen Failure
Description: The time to prostate specific antigen failure was defined as the days from first dosing (scheduled dosing days) where an increase in serum prostate specific antigen of ≥50% from nadir and a least 5 ng/mL measured on two consecutive occasions at least two weeks apart was noted.
Time Frame: 12 months
Population: ITT population. Missing values were not imputed for this endpoint. Number in table represents the number of patients with prostate-specific antigen failure.
Measure: Number; unit: participants
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
participants
  Day 0-28 (patients at risk=193, 201, 194) | 1 | 0 | 1
  Day 0-56 (patients at risk=192, 197, 192) | 1 | 0 | 1
  Day 0-84 (patients at risk=190, 193, 190) | 1 | 0 | 1
  Day 0-112 (patients at risk=190, 189, 188) | 1 | 1 | 3
  Day 0-140 (patients at risk=187, 187, 182) | 2 | 2 | 7
  Day 0-168 (patients at risk=179, 185, 180) | 7 | 4 | 9
  Day 0-196 (patients at risk=173, 181, 175) | 11 | 4 | 11
  Day 0-224 (patients at risk=168, 175, 173) | 14 | 7 | 12
  Day 0-252 (patients at risk=165, 169, 168) | 16 | 9 | 14
  Day 0-280 (patients at risk=157, 165, 163) | 20 | 11 | 18
  Day 0-308 (patients at risk=153, 161, 156) | 23 | 12 | 21
  Day 0-336 (patients at risk=149, 156, 150) | 26 | 15 | 24
  Day 0-364 (patients at risk=149, 155, 148) | 26 | 16 | 26
Statistical Analysis 1: Comparison: Degarelix 240/160 mg; Test type: Superiority or Other; Cumulative probability = 85.8, 95% CI [79.8 to 90.1] — 95% confidence interval for the cumulative probability of completing the study without prostate specific antigen failure from Day 0 to Day 364
Statistical Analysis 2: Comparison: Degarelix 240/80 mg; Test type: Superiority or Other; Cumulative probability = 91.1, 95% CI [85.9 to 94.5] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Leuprolide 7.5 mg; Test type: Superiority or Other; Cumulative probability = 85.9, 95% CI [79.9 to 90.2] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Participants With Markedly Abnormal Change in Laboratory Variables (>=20 Percent of Patients)
Description: Criteria for lab values changes from baseline to the end of the study considered markedly abnormal were set for each lab test. If 20% of patients reached that value, the results were reported.
Time Frame: Baseline to Day 364
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
participants
  Haematocrit (<=0.37 ratio) | 73 | 80 | 73
  Haemoglobin (<=115 g/L) | 32 | 45 | 38
  Serum Urea Nitrogen (>=10.7 mmol/L) | 48 | 41 | 50
  Urine Protein (>=2 units from baseline) | 65 | 64 | 63
  Urine Bacteria (0 at baseline and >0 on treatment) | 96 | 105 | 107

8. Secondary Outcome: The Mean Value of QTc Interval as Measured by Electrocardiogram
Description: The QTc interval results are calculated with Fridericia's correction. QTc intervals are a standard evaluation of an electrocardiogram and help measure the risk of developing ventricular arrhythmias.
Time Frame: 12 months
Population: ITT population. End of Study values obtained at day 364 (+-7 days) for patients who completed. Patients who withdrew early had variable timeframes for the end of study value.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
milliseconds
  Baseline Day 0 (n=202, 207, 201) | 403 (20.2) | 407 (21.6) | 404 (19.4)
  Day 3 (n=195, 204, 197) | 404 (22.1) | 411 (23.5) | 405 (23.0)
  End of study 12 months (n=202, 207, 201) | 415 (21.7) | 420 (22.3) | 419 (23.3)

9. Secondary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: Vital signs and body weight included incidence of markedly abnormal changes from baseline to the end of the study in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of patients in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 12 months
Population: ITT population. The first value in the category represents the actual clinical reading and the second is the change from baseline for blood pressure (units: millimeters of mercury) and heart rate (units:beats per minute). The weight category includes patients whose percent weight change from baseline fit the stated ranges.
Measure: Number; unit: participants
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Number analyzed (Participants) | 202 | 207 | 201
participants
  Systolic blood pressure <=90 and decrease >=20 | 12 | 8 | 6
  Systolic blood pressure >=180 and increase >=20 | 20 | 16 | 23
  Diastolic blood pressure <=50 and decrease >=15 | 12 | 10 | 9
  Diastolic blood pressure >=105 and increase >=15 | 5 | 13 | 8
  Heart rate <=50 and decrease >=15 | 8 | 7 | 9
  Heart rate >=120 and increase >=15 | 1 | 0 | 1
  Body weight decrease of >=7 percent | 5 | 6 | 10
  Body weight increase of >=7 percent | 24 | 15 | 23

ADVERSE EVENTS:
Arm/Group | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Serious Adverse Events (participants affected / at risk) | 24 | 21 | 28
Other Adverse Events (participants affected / at risk) | 165 | 162 | 153
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Anaemia (Blood and lymphatic system disorders) | 2/202 (2) | 0/207 (0) | 3/201 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Cardiac arrest (Cardiac disorders) | 0/202 (0) | 2/207 (2) | 0/201 (0)
Acute coronary syndrome (Cardiac disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Acute myocardial infarction (Cardiac disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Angina unstable (Cardiac disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Bradycardia (Cardiac disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Cardiac failure (Cardiac disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Cardiopulmonary failure (Cardiac disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Coronary artery disease (Cardiac disorders) | 0/202 (0) | 1/207 (1) | 1/201 (1)
Myocardial infarction (Cardiac disorders) | 0/202 (0) | 1/207 (1) | 2/201 (2)
Cardiac disorder (Cardiac disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Cardiac failure congestive (Cardiac disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Cardiovascular disorder (Cardiac disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Myocardial ischaemia (Cardiac disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Myopericarditis (Cardiac disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Cataract (Eye disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Inguinal hernia (Gastrointestinal disorders) | 1/202 (1) | 1/207 (1) | 0/201 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Gastritis (Gastrointestinal disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Peritonitis (Gastrointestinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Non-cardiac chest pain (General disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Pyrexia (General disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Hepatic failure (Hepatobiliary disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Hepatomegaly (Hepatobiliary disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Bronchopneumonia (Infections and infestations) | 1/202 (1) | 1/207 (1) | 0/201 (0)
Ear infection (Infections and infestations) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Gastroenteritis (Infections and infestations) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Lobar pneumonia (Infections and infestations) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Pneumonia (Infections and infestations) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Post procedural cellulitis (Infections and infestations) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Overdose (Injury, poisoning and procedural complications) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Prostate examination abnormal (Investigations) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Blood creatinine increased (Investigations) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Electrocardiogram (ECG) signs of myocardial ischaemia (Investigations) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Dehydration (Metabolism and nutrition disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/202 (1) | 1/207 (1) | 1/201 (1)
Malignant lymphoma unclassifiable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Linitis plastica (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Cerebral infarction (Nervous system disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Cerebrovascular accident (Nervous system disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Hyperkinesia (Nervous system disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Syncope (Nervous system disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Haematuria (Renal and urinary disorders) | 2/202 (2) | 1/207 (1) | 0/201 (0)
Calculus bladder (Renal and urinary disorders) | 1/202 (1) | 1/207 (1) | 0/201 (0)
Calculus ureteric (Renal and urinary disorders) | 0/202 (0) | 2/207 (2) | 1/201 (1)
Urinary retention (Renal and urinary disorders) | 2/202 (2) | 0/207 (0) | 2/201 (2)
Bladder obstruction (Renal and urinary disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Hydronephrosis (Renal and urinary disorders) | 1/202 (2) | 0/207 (0) | 1/201 (1)
Renal failure acute (Renal and urinary disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Renal failure chronic (Renal and urinary disorders) | 1/202 (2) | 0/207 (0) | 0/201 (0)
Urethral obstruction (Renal and urinary disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Renal failure (Renal and urinary disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Urethral stenosis (Renal and urinary disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/202 (1) | 0/207 (0) | 0/201 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0/202 (0) | 0/207 (0) | 1/201 (1)
Hypertension (Vascular disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Hypotension (Vascular disorders) | 0/202 (0) | 1/207 (1) | 0/201 (0)
Orthostatic hypotension (Vascular disorders) | 1/202 (1) | 0/207 (0) | 1/201 (1)
Deep vein thrombosis (Vascular disorders) | 0/202 (0) | 0/207 (0) | 2/201 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 240/160 mg | Degarelix 240/80 mg | Leuprolide 7.5 mg
Nausea (Gastrointestinal disorders) | 11/202 (15) | 9/207 (10) | 8/201 (9)
Constipation (Gastrointestinal disorders) | 6/202 (6) | 11/207 (12) | 10/201 (11)
Injection site pain (General disorders) | 61/202 (108) | 58/207 (114) | 1/201 (1)
Injection site erythema (General disorders) | 48/202 (63) | 36/207 (56) | 0/201 (0)
Injection site swelling (General disorders) | 14/202 (23) | 13/207 (17) | 0/201 (0)
Fatigue (General disorders) | 13/202 (14) | 7/207 (11) | 13/201 (14)
Injection site induration (General disorders) | 11/202 (14) | 8/207 (11) | 0/201 (0)
Injection site nodule (General disorders) | 13/202 (24) | 6/207 (8) | 0/201 (0)
Chills (General disorders) | 7/202 (9) | 11/207 (19) | 0/201 (0)
Urinary tract infection (Infections and infestations) | 3/202 (3) | 10/207 (14) | 18/201 (25)
Weight increased (Investigations) | 22/202 (22) | 18/207 (18) | 24/201 (24)
Alanine aminotransferase increased (Investigations) | 17/202 (17) | 20/207 (22) | 11/201 (11)
Aspartate aminostransferase increased (Investigations) | 10/202 (11) | 11/207 (12) | 6/201 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12/202 (12) | 7/207 (7) | 5/201 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 12/202 (13) | 12/207 (12) | 17/201 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6/202 (6) | 11/207 (12) | 18/201 (20)
Hot flush (Vascular disorders) | 53/202 (59) | 53/207 (71) | 43/201 (50)
Hypertension (Vascular disorders) | 14/202 (16) | 11/207 (12) | 8/201 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.